CLINICAL TRIAL: NCT06477354
Title: ACEMg (Soundbites) Hearing Preservation, Tinnitus and Hyperacusis Relief Otology Intervention Study
Brief Title: ACEMg Hearing Preservation, Tinnitus and Hyperacusis Relief
Acronym: OTISRWD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keep Hearing, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ACEMg OTIS Study
Record Dates: First submitted 2024-06-05; First posted 2024-06-27 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Sensorineural Hearing Loss; Tinnitus; SNHL; Inner Ear Hearing Loss
Keywords: Phase IV open-label post-marketing surveillance; Hearing preservation; Tinnitus; SNHL; Hearing preventive care; ACEMg; Nutraceutical; Real-world data (RWD) analysis; Soundbites; Tinnitus symptom refief
MeSH Terms: conditions — Hearing Loss, Sensorineural; Tinnitus

STUDY DESIGN:
Intervention Model Description: Open-label, post-marketing surveillance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- At-home (Experimental): Subjective auditory function assessments with the hearWHO app. Tinnitus survey. Participants take ACEMg softgel capsules daily, self-administered orally.
  Interventions: Dietary Supplement: ACEMg

INTERVENTIONS:
Dietary Supplement: ACEMg — Softgel capsules
  Other Names: Soundbites

SUMMARY:
ACEMg (Soundbites) is a neuroprotectant supplement designed to block the initiating biological events in the inner ear leading to inner ear hearing loss, sensorineural hearing loss, SNHL, which accounts for more than 90% of all hearing loss. SNHL is so common it is called hearing loss. There is no cure for SNHL.

The 24-week OTIS Study aims to validate findings from the previous two-year real-world study demonstrating ACEMg (Soundbites) preserved or improved auditory function (hearing) for 75.3% of participants who used it daily, with most improvement occurring within six months.

The study also aims to assess the potential of ACEMg to relieve tinnitus, hyperacusis, and hearing sensitivity symptoms. These symptoms are often correlated with SNHL; relief from tinnitus, hyperacusis and hearing sensitivity were were not measured in the previous two-year study.

The OTIS study aims to answer two questions. First, does the real-world data demonstrate that hearing loss is stabilized or improved at the end of the test among participants with SNHL at the beginning? Second, do participants who self-report tinnitus, hyperacusis, or hearing sensitivity symptoms at the start of their test report reduced symptoms at the end?

Participants must be eighteen years of age and older and self-report hearing loss and/or tinnitus. The study is conducted at home using a smartphone app and a web-based assessment and data reporting tool developed for this study.

The study is conducted at home using an online hearing test and short surveys on tinnitus and hyperacusis. The tests are completed three times: Baseline tests are taken before participants begin to take ACEMg softgel capsules daily. The Test is repeated at about 11 and 24 weeks. Assessment scores at the beginning of the study will be compared with scores at the end.

Participation in the study is free.

DETAILED DESCRIPTION:
OVERVIEW

The 2-year Soundbites Real World Evidence study used otoacoustic emissions examinations conducted by an audiologist to assess auditory function objectively. Soundbites was clinically proven to preserve or improve hearing for 75.3% of those who took it daily. Among those who benefited, hearing loss stopped for half and improved for the other half. Most of the benefits happened within the first 6 months. Results continued with ongoing use.

ACEMg and tinnitus

ACEMg was not designed to address tinnitus or hyperacusis, and the 2-year study did not assess either. Nevertheless, since ACEMg became available as Soundbites softgel capsules in 2017, reports from customers with tinnitus and from audiologists treating patients with tinnitus or hyperacusis indicate that ongoing daily use of Soundbites relieves tinnitus and hyperacusis symptoms for some.

Assessing ACEMg for tinnitus symptom relief

An effective cure for tinnitus does not exist, and hyperacusis and tinnitus symptoms are correlated. However, research indicates that often, the initial step in tinnitus development is damage to outer hair cells in the cochlea, precisely what ACEMg is designed to block.

That is the rationale for including tinnitus assessments in this follow-on OTIS Study. Many studies aim to reduce the cognitive impacts of permanent, chronic tinnitus by employing various brain training techniques. The OTIS Study is believed to be the first aiming to assess the potential of a clinically proven inner ear neuroprotectant to relieve tinnitus symptoms directly. We hypothesize that a cochlear neuroprotectant intervention may relieve tinnitus symptoms for some.

Who can participate?

The study is open to those eighteen years and older who self-report hearing loss and/or tinnitus and have not used ACEMg as Soundbites.

How the study works.

The OTIS Study is a collaboration between Keep Hearing Initiative (Keep Hearing), the study sponsor, and Soundbites Public Benefit Corporation (Soundbites PBC). Keep Hearing is responsible for IRB compliance, data analysis, and public health reporting. Soundbites PBC donates the ACEMg test product and is responsible for data collection. Both partners are responsible for recruitment, enrollment, and data security.

Participants conduct the study at home and report their data online using a secure, automated web-based tool developed specifically for the OTIS Study by Soundbites Public Benefit Corporation, the maker of ACEMg as Soundbites softgel capsules.

BACKGROUND OF THE INTERVENTION

ACEMg, developed at the University of Michigan Medical School, is designed to block the initiating biochemical events in the organ of Corti within the inner ear leading to sensorineural hearing loss (SNHL).

The ACEMg formula is classified as Generally Regarded as Safe (GRAS) by the U.S. Pharmacopeia and regulated as a dietary supplement under FDA DSHEA law. The ACEMg patents are licensed to Soundbites Public Benefit Corporation (PBC), which produces an updated and improved oral softgel capsule dose format of ACEMg for adults, and an oral twist-off softgel capsule format for children, available to the public without a prescription under the Soundbites trademark.

PREVIOUS REAL-WORLD EVIDENCE RESEARCH

The 2021-2023 ACEMg (Soundbites) Real-world Evidence Study (N=190) used de-identified real-world data (RWD) from routine annual otoacoustic emissions (OAE) examinations collected among adult patients of one audiology practice over many years before ACEMg became available. OAE examinations produce objective measures of inner ear auditory function.

The control dataset (N=97) represented the current standard of care for hearing, which is to say no treatment. Retrospective OAE RWD from the no-treatment group was analyzed and compared to RWD from a treatment group of patients (N=93) who also had at least two years of annual retrospective OAE examinations and began taking ACEMg immediately following their third annual OAE examination, thus enabling objective measurement of the potential impacts on auditory function from daily oral self-administration of ACEMg.

The study yielded statistically significant clinical data demonstrating that ACEMg effectively preserved and improved auditory function, thereby mitigating SNHL, demonstrating that ACEMg preserved or improved inner ear auditory function for 75.3% (N=70) of those in the treatment group (N=93), with most improvement occurring within the first six months of daily use.

The article reporting results from the study is available on the Open Science Framework (OSF) preprint server at https://osf.io/preprints/osf/uw7tq.

Study administrators concluded that the clinical data justify a larger study, especially considering the inherent safety of ACEMg and its availability in an inexpensive, convenient oral dose form, perhaps leading to considering ACEMg as an effective, accessible method of addressing the global public health challenge of hearing loss.

OTIS STUDY Inclusion and exclusion criteria

Individuals eighteen years or older and self-report hearing loss and/or tinnitus may participate. A personal email account and U.S. mailing address are required.

Individuals younger than eighteen years, those who do not have hearing loss or tinnitus, those who have previously taken Soundbites, and those who cannot take the micronutrients beta carotene, vitamin C, vitamin E or Magnesium are excluded from participating.

Method

All potential participants download, read, review, and discuss the informed consent and data-sharing agreement with the study coordinator. Participants accept the agreement online and begin testing ACEMg as Soundbites softgel capsules at home for 24 weeks about 6 months.

The test starts with a baseline hearing assessment of hearing with the hearWHO digits-in-hearing app developed for the World Health Organization until remote otoacoustic emissions (OAE) test technology becomes available.

The hearWHO app is available free to the general public. It is recommended for people who listen to loud music over personal audio devices and can also be used by health workers to screen people for hearing loss. The app is intended for use by people 18 years of age and above and may not provide reliable results for children.

Participants self-reporting tinnitus symptoms complete the tinnitus survey which uses questions selected from the Tinnitus Handicap Inventory to assess the degree to which tinnitus symptoms impact daily activities.

All participant data is private. Data is entered into a private, passcode-protected online tool developed for the study. Data is stored on the Open Science Framework online data store. Collected data is limited to birth date, gender, assessment dates, and assessment scores. Participants record their baseline test scores before starting to take ACEMg as Soundbites softgel capsules for adults daily. The hearing test and/or tinnitus survey are repeated at about 12 and 24 weeks.

Data sharing, analysis and reporting

By accepting the terms of the informed consent and data-sharing agreement upon joining the study, participants agree to submit their de-identified data for analysis and reporting after their 24-week test is complete. All data is shared for secondary analysis and reporting under a data-sharing agreement with the study sponsor, the Keep Hearing nonprofit.

Analysis of each participant's results is shared with each participant immediately upon completion of their individual 24-week study. Aggregated data analyses will be reported in publicly available manuscripts submitted for peer review.

Costs

Participation in the study is free. Soundbites Public Benefit Corporation donates the Soundbites softgel capsules, U.S. delivery costs, and the online data entry and data storage tool.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus self-reported at the baseline survey, or
* Hearing loss assessed at the baseline test

Exclusion Criteria:

* No tinnitus self-reported at the baseline survey, or
* No hearing loss assessed at the baseline test
* Previous use of ACEMg (Soundbites)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Subjective measure of preservation or improvement of inner ear auditory function | Time point zero; 12 and 24 weeks.
  Hearing assessments using the hearWHO digits-in-noise test
Tinnitus symptom relief | Time point zero; 12 and 24 weeks.
  Subjective assessment of tinnitus symptoms using the tinnitus survey

CONTACTS AND LOCATIONS:
Overall Officials: Barry Seifer, MFA, Study Director — Keep Hearing, Inc. 501c3
Locations (1):
- To enroll, visit the Participate in Public Health Research page on keephearing.org, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Impact of the ACEMg Biomedicine on Sensorineural Hearing Loss and Auditory Function: Analysis of Real-World Clinical Data — https://osf.io/preprints/osf/uw7tq